CLINICAL TRIAL: NCT01142804
Title: WalkLink:Internet-based Walking Program for Cardiovascular Disease Risk-Reduction
Brief Title: WalkLink: Internet-based Walking Program
Acronym: WalkLink
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Liza Rovniak, Assistant Professor of Medicine and Public Health Sciences, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IRB-31708
Record Dates: First submitted 2010-06-10; First posted 2010-06-11 (Estimated); Last update posted 2015-08-13 (Estimated); Status verified 2015-08

CONDITIONS: Physical Activity
Keywords: Walking programs; Physical Activity; Behavior Modification; Social Support
MeSH Terms: conditions — Motor Activity | interventions — Population Groups

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Enhanced Usual Care Group (Experimental): Participants received weekly emailed tips of the week to provide support for walking.
  Interventions: Behavioral: Group
- WalkLink Group (Experimental): Participants received weekly emailed tips of the week, plus evidence-based online fitness walking program.
  Interventions: Behavioral: Group
- WalkLink+ Group (Experimental): Participants received weekly emailed tips, plus evidence-based online fitness walking program, plus online/in-person social network intervention.
  Interventions: Behavioral: Group

INTERVENTIONS:
Behavioral: Group — Walking programs with various levels of support will be administered to determine which one is most effective.
  Other Names: Enhanced Usual Care; WalkLink; WalkLink+

SUMMARY:
The investigators propose a randomized controlled trial based on the Social Networks for Activity (SNAP) Model to evaluate: (1) the effectiveness of an internet-based fitness walking program delivered to patients with risk factors for cardiovascular disease and stroke; and (2) the contribution of social support networks to enhancing the effectiveness of the internet-based fitness walking program. The investigators will recruit 308 patients who are sedentary and have risk factors for cardiovascular disease and randomly assign them to one of the following groups: 1. Internet-based fitness walking program (WalkLink); 2. Internet-based fitness walking program plus additional social network intervention (WalkLink+); and 3. Minimal treatment control.

The primary specific aims of this study are to:

1. Evaluate the effects of WalkLink and WalkLink+ relative to a minimal treatment control group on change in: physical activity, aerobic fitness, blood pressure, body composition, and body mass index (BMI), from baseline to posttest, and at 6-month follow-up.
2. Compare the differential effectiveness of WalkLink+ to WalkLink on change in: physical activity, aerobic fitness, blood pressure, body composition and BMI from baseline to posttest, and at 6-month follow-up.
3. Evaluate the mediator and moderator effects of selected individual-level self-management skills (goal setting, planning, self-monitoring), social support variables (number of activity partners, social cues for walking, social praise/reinforcement), and physical-ecological variables (neighborhood walkability, physical cues for walking) on WalkLink and WalkLink+ treatment outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Sedentary, defined as less than 150 minutes per week of moderate intensity activity
* Between the ages of 35 and 64
* Able to speak English
* Able to provide informed consent
* Able to participate in moderate-intensity physical activity (e.g., moderate pace walking)

Exclusion Criteria:

* No access to home or private work computer with Internet access
* Body mass index (BMI) greater than 39.9
* Systolic blood pressure > 160 mm Hg or diastolic blood pressure > 100 mm Hg
* Bone, joint, or foot problems that interfere with walking
* Diabetes, pulmonary, or cardiovascular disease
* Consume 5 or more drinks of alcohol a day
* Currently pregnant
* Not living within the preselected study neighborhoods or plan to move from the local area during the study period

Ages: 35 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 308 (Actual)
Dates: Start 2010-08; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Moderate Vigorous Activity | 9 months
  Change in Moderate Vigorous Activity will be assessed using Actigraph accelerometers

SECONDARY OUTCOMES:
Health Risk Factors | 9 months
  Aerobic fitness, blood pressure, body mass index, body composition

OTHER OUTCOMES:
Environmental Factors | 9 months
  Built and social environment factors

CONTACTS AND LOCATIONS:
Overall Officials: Liza Rovniak, PhD, MPH, Principal Investigator — Penn State College of Medicine, Penn State Milton S. Hershey Medical Center
Locations (1):
- Penn State College of Medicine, Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania, United States

REFERENCES:
- [Derived] Rovniak LS, Kong L, Hovell MF, Ding D, Sallis JF, Ray CA, Kraschnewski JL, Matthews SA, Kiser E, Chinchilli VM, George DR, Sciamanna CN. Engineering Online and In-Person Social Networks for Physical Activity: A Randomized Trial. Ann Behav Med. 2016 Dec;50(6):885-897. doi: 10.1007/s12160-016-9814-8. PMID 27405724
- [Derived] Rovniak LS, Sallis JF, Kraschnewski JL, Sciamanna CN, Kiser EJ, Ray CA, Chinchilli VM, Ding D, Matthews SA, Bopp M, George DR, Hovell MF. Engineering online and in-person social networks to sustain physical activity: application of a conceptual model. BMC Public Health. 2013 Aug 14;13:753. doi: 10.1186/1471-2458-13-753. PMID 23945138